CLINICAL TRIAL: NCT03366883
Title: A Phase III Trial Comparing Paclitaxel, Cisplatin Plus 5-FU (TCF) Versus Radiotherapy With Paclitaxel Plus Cisplatin (TC-RT) as Preoperative Therapy for Locally Advanced Esophageal Squamous Cancer
Brief Title: Paclitaxel, Cisplatin,5-FU vs. Radiotherapy Plus Paclitaxel, Cisplatin as Preoperative Therapy for Locally Advanced ESC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Shanghai Chest Hospital (Other); Henan Cancer Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); First Affiliated Hospital of Chongqing Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TianjinCIH20171114
Record Dates: First submitted 2017-11-14; First posted 2017-12-08 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-11

CONDITIONS: Esophageal Cancer Stage IIB; Esophageal Cancer Stage III
Keywords: preoperative chemotherapy; preoperative chemoradiotherapy; clinical trial; phase III; Esophageal squamous cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Cisplatin; Fluorouracil; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Paclitaxel, Cisplatin Plus 5-FU (TCF) (Experimental): preoperative chemotherapy with three cycles of TCF(Paclitaxel 135mg/m2 D1;Cisplatin 60mg/m2 D1 or 20mg/m2 D1-D3;5-fluorouracil 600mg/m2 D1-D5；repeated every 3 weeks
  Interventions: Combination Product: Paclitaxel, Cisplatin Plus 5-FU (TCF)
- Preoperative radiochemotherapy (Experimental): preoperative radiochemotherapy (41.4 Gy/23 fractions or 40 Gy/20 fractions) with four cycles of TP(Paclitaxel 45mg/m2 on D1 and Cisplatin 20mg/m2 D1,repeated every week
  Interventions: Radiation: radiochemotherapy

INTERVENTIONS:
Combination Product: Paclitaxel, Cisplatin Plus 5-FU (TCF) — preoperative chemotherapy with three cycles of TCF(Paclitaxel 135mg/m2 D1;Cisplatin 60mg/m2 D1 or 20mg/m2 D1-D3;5-fluorouracil 600mg/m2 D1-D5；repeated every 3 weeks)
  Arms: "Paclitaxel, Cisplatin Plus 5-FU (TCF)
Radiation: radiochemotherapy — preoperative radiochemotherapy (41.4 Gy/23 fractions or 40 Gy/20 fractions) with four cycles of TP(Paclitaxel 45mg/m2 on D1 and Cisplatin 20mg/m2 D1,repeated every week)
  Arms: Preoperative radiochemotherapy

SUMMARY:
This is a Phase III clinical trail which Comparing Paclitaxel, Cisplatin Plus 5-FU (TCF) Versus Radiotherapy with Paclitaxel Plus Cisplatin (TC-RT) as Preoperative Therapy for Locally Advanced Esophageal Squamous Cancer. The Preoperative chemoradiotherapy with radical surgery is the standard treatment in China. But, many patients do not receive this treatment for many other reasons. Most of them refused or abandon radiotherapy because of the Intolerable adverse effects of radiotherapy, so we have launched a randomized controlled trial to confirm the non-inferiority of TCF over chemoradiotherapy with TC (TC-RT) as preoperative therapy for locally advanced esophageal squamous cancer in overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma.
* All lesions are located in the thoracic esophagus.
* Clinical stages IIB and III (excluding T4) based on the 7th UICC-TNM classification.
* 20-75 years old.
* ECOG performance status of 0 or 1.
* Measurable lesions not required.
* No prior therapy against esophageal cancer except for complete resection by endoscopic mucosal resection/endoscopic submucosal dissection with either pM1/M2 disease or pM3 disease without vascular infiltration.
* No prior chemotherapy, radiotherapy or hormonal therapy against any cancers
* Adequate organ function.
* Written informed consent.

Exclusion Criteria:

* Synchronous or metachronous double cancers, except for intramucosal tumor curatively resected by local therapy.
* Active infection requiring systemic therapy
* Positive hepatitis B surface antigen and hepatitis B core antigen or human immunodeficiency virus antibody.(only positive hepatitis B surface antigen should receive anti-virus treatment during study)
* Pregnant or lactating women or women of childbearing potential.
* Patients requiring systemic steroid medication.
* Iodine hypersensitivity.
* Psychiatric disease.
* Hypersensitivity for CremophorEL.
* Poorly controlled diabetes.
* Severe emphysema or pulmonary fibrosis.
* Poorly controlled hypertension.
* Unstable angina within 3 weeks or with a history of myocardial infarction within 6 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2018-02-04 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years

SECONDARY OUTCOMES:
Disease Free Survival | 3years
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average of 1 year
  All participants with treatment-related adverse events as assessed by CTCAE v4.0
Objective Response Rate | up to 24 weeks
Rate of R0 resection | up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- TianjinCIH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No